CLINICAL TRIAL: NCT01023113
Title: To Compare Visual Field Impairment in Conventional Double Frequency Nd: YAG Panretinal Photocoagulation With PASCAL Panretinal Photocoagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: LVPrasad Eye Institute Hyderabad, Same as above
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nand2010
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Macular Edema; Diabetic Retinopathy; Visual Field Loss
Keywords: Diabetic retinopathy; laser; field loss; macular edema; Visual field loss
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PASCAL laser, PRP in 2-3 sitting at 3 days interval. (Experimental): PRP will be completed in 2-3 sitting at 3 days interval with one spots apart and moderate intensity gray burns will be given between arcade to periphery by PASCAL laser
  Interventions: Procedure: PASCAL laser
- Conventional laser (Active Comparator): PRP will be completed in 2-3 sitting at 3 days interval with one spots apart and moderate intensity gray burns will be given between arcade to periphery by conventional laser
  Interventions: Procedure: Conventional laser

INTERVENTIONS:
Procedure: PASCAL laser — PRP will be completed in 2-3 sitting at 3 days interval with one spots apart and moderate intensity gray burns will be given between arcade to periphery
  Arms: PASCAL laser, PRP in 2-3 sitting at 3 days interval.
Procedure: Conventional laser — PRP will be completed in 2-3 sitting at 3 days interval with one spots apart and moderate intensity gray burns will be given between arcade to periphery
  Arms: Conventional laser

SUMMARY:
Lacunae in Knowledge No study is available in literature regarding visual field impairment in proliferative diabetic retinopathy comparing conventional double frequency Nd:YAG panretinal photocoagulation with PASCAL panretinal photocoagulation

AIMS & OBJECTIVE

1. To compare visual field impairment in conventional double frequency Nd: YAG panretinal photocoagulation with PASCAL panretinal photocoagulation.
2. To examine the effect of these modalities of laser on macular edema

60 eyes of proliferative diabetic retinopathy will undergo humphery visual field analysis,and optical coherence tomography before and after panretinal photocoagulation

DETAILED DESCRIPTION:
Material and Methods

1.Study will be prospective randomized interventional case series. Methods: 60 eyes of proliferative diabetic retinopathy (clear media with no vitreous/significant preretinal hemorrhage) will be taken for the study, out of which 30 eyes will undergo panretinal photocoagulation by conventional frequency doubled Nd: YAG laser and remaining 30 eyes will be by PASCAL laser.

All patients will undergo routine ophthalmic examination (visual acuity, slit lamp, indirect ophthalmoscope, IOP) as well as FFA/seven fields fundus photos (whenever required), OCT(optoview spectral domain OCT), visual fields (Humphrey 30-2 SITA Standard and 60-1) and baseline blood investigation will be done before 1st sitting of laser. Written informed consent will be taken by all the subjects. PRP will be completed in 2-3 sitting at 3 days interval with one spots apart and moderate intensity gray burns will be given between arcade to periphery. In case of clinical significant macular edema modified grid/ focal laser of mild intensity spots will be done. At each visit patient will be assessed for visual acuity, OCT, IOP (applanation tonometer). Patients will be followed up for at least 3 months. After the completion of last sitting of photocoagulation, follow-up will be at one month and 3 months. At one month follow up together with routine ophthalmic examination, OCT, HVF 30-2,60-1 will be done. At final follow-up at 3 months HVF 30-2,60-1,OCT will be done in addition of routine ophthalmic examination and FFA will be done whenever indicated.

Inclusion Criteria

1. 60 eyes of diabetic patients with proliferative DR will be included.
2. Visual acuity 20/50 or better in all patients.
3. Patients available for follow up at least twice between 4-12 weeks.
4. Patients giving consent for panretinal photocoagulation and for inclusion in study

Exclusion Criteria

1. Patients with diseases known to affect visual ﬁeld as such as aphakia, cataract, glaucoma, optic nerve and macular diseases, will be excluded from the study.
2. Previous photocoagulation(macular laser or PRP) will also be an exclusion criterion.

Out come Measure

1. Comparison of the two methods in relation to visual field loss(in previous studies average deterioration in visual field(MD) was 3-5dB in 45% cases) in terms of MD,CPSD and each quadrants loss of fields and number of patients worsened the visual fields and which method will be superior in term of less visual field loss.
2. Effect on macular edema in terms of OCT thickness

ELIGIBILITY:
Inclusion Criteria:

1. 60 eyes of diabetic patients with proliferative DR will be included.
2. Visual acuity 20/50 or better in all patients.
3. Patients available for follow up at least twice between 4-12 weeks.
4. Patients giving consent for panretinal photocoagulation and for inclusion in study

Exclusion Criteria:

1. Patients with diseases known to affect visual ﬁeld as such as aphakia, cataract, glaucoma, optic nerve and macular diseases, will be excluded from the study.
2. Previous photocoagulation(macular laser or PRP) will also be an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of the two methods in relation to visual field loss in terms of MD,CPSD and each quadrants loss of fields | 3 months

SECONDARY OUTCOMES:
Effect on macular edema in terms of OCT thickness | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- LV Prasad Eye Institute, Hyderabad, A.P., India